CLINICAL TRIAL: NCT01687426
Title: A Single-Center, Randomized, Double-Masked, Cross-Over Pilot Study Evaluating Safety and IOP Lowering Response of Brimonidine Tartrate Ophthalmic Solution Versus Vehicle in Subjects With Open Angle Glaucoma or Ocular Hypertension
Brief Title: Study Evaluating the Safety and Intraocular Pressure (IOP) Lowering Response of Brimonidine Tartrate Ophthalmic Solution in Subjects With Open Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eye Therapies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 12-150-0001
Record Dates: First submitted 2012-09-05; First posted 2012-09-19 (Estimated); Last update posted 2012-12-25 (Estimated); Status verified 2012-12

CONDITIONS: Glaucoma and Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brimonidine Tartrate 0.025% (Active Comparator)
  Interventions: Drug: Brimonidine Tartrate 0.025%; Drug: Vehicle
- Vehicle (Placebo Comparator)
  Interventions: Drug: Brimonidine Tartrate 0.025%; Drug: Vehicle

INTERVENTIONS:
Drug: Brimonidine Tartrate 0.025% — 1 drop in each eye daily four times a day for 14 days
Drug: Vehicle — 1 drop in each eye daily four times a day for 14 days

SUMMARY:
The purpose of this study is to determine the intraocular Pressure (IOP) lowering response and evaluate the safety of brimonidine tartrate 0.025% ophthalmic solution in adult subjects with open angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age at Visit 1 (Screening), of either sex and any race
* Be willing and able to provide written informed consent prior to any study procedures being performed.
* Be willing and able to follow all instructions and attend all study visits.
* Be willing to discontinue use of disallowed medication
* Have a documented diagnosis of ocular hypertension, open angle glaucoma or chronic angle closure glaucoma with a patent iridotomy.

Exclusion Criteria:

* Have known sensitivity or poor tolerance to brimonidine or any other component of the study medications.
* Have any form of glaucoma other than open-angle glaucoma, ocular hypertension or chronic angle closure glaucoma with patent iridotomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
IOP | 14 days

OTHER OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety | For up to 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Site, Winchester, Massachusetts, United States